CLINICAL TRIAL: NCT07299721
Title: Brain Ultrafast Ultrasound Imaging: Application in Pediatric Cardiology: Brain Ultrafast
Brief Title: Brain Ultrafast Ultrasound Imaging
Acronym: Brain Ultrafas
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2025/28; CER-BDX 2025-136 (Other: Comité d'Etique - Centre Ethique et Recherche en Santé de Bordeaux)
Record Dates: First submitted 2025-11-19; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: CHD - Congenital Heart Disease
Keywords: Congenital Heart Disease; Paediatric; Cardiac Imaging; Ultrafast ultrasounf
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient receiving a transcranial Doppler: Every patient receiving a transcranial Doppler in routine care in our CHD unit of intensive care and anaesthesiology for cardiovascular surgery department
  Interventions: Other: Ultrafast ultrasound (UFUS)

INTERVENTIONS:
Other: Ultrafast ultrasound (UFUS) — Ultrafast ultrasound imaging(UFUS), ultrasound images at a very high rate, using a Verasonics system (ultrasound open platform).

SUMMARY:
Congenital heart defects affect 1 in 100 births in France, with rising prevalence due to better care. Despite improved survival, 40% of children post-surgery face neurological impairments, and some of them show brain lesions. Causes include heart defects, genetic syndromes, and surgeries. Some heart defects and support systems increase cerebral risks. Monitoring cerebral perfusion is difficult to assess but emerging ultrafast ultrasound offers real-time, non-invasive blood flow insights.

DETAILED DESCRIPTION:
Congenital heart defects affect 1 in 100 live births in France. While incidence remains stable, prevalence is rising due to improved medical care, with cases expected to double by 2050. Despite increased survival, neurological comorbidities remain a major concern, with 40% of patients undergoing childhood cardiac surgery experiencing impairments and 73% presenting MRI-detectable brain lesions postoperatively. These injuries result from congenital heart defects, haemodynamic disturbances, genetic syndromes, and neonatal surgeries with extracorporeal circulation.

Some heart defects, such as systemic-to-pulmonary shunts and cyanotic heart diseases, impair cerebral perfusion, increasing the risk of hypoxia and stroke. Mechanical circulatory support systems (e.g. ECMO, cardiopulmonary bypass) also contribute to cerebral risks due to hypoperfusion and clotting complications.

Cerebral autoregulation helps maintain stable perfusion despite blood pressure variations. However, bedside cerebral perfusion monitoring remains challenging leading to reliance on indirect methods like near-infrared spectroscopy (NIRS) and transcranial Doppler (TCD), both with limitations. Ultrafast ultrasound (UFUS) is an emerging non-invasive technique that enables real-time quantification of cerebral blood flow, offering new insights into neonatal cerebral haemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Every patient under 2 years old any sex or gender hospitalised in the congenital heart disease unit of the intensive care and anaesthesia for cardiovascular surgery, CHU de Bordeaux.
* Open anterior fontanella
* congenital heart disease
* cardiac shock necessitating mechanical circulatory support.
* Social security affiliation
* Parental or legal guardian's non-opposition

Exclusion Criteria:

* Anechoic
* Allergy to echocardiography gel.

Ages: 0 Years to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Every patient, under two years old, receiving a transcranial Doppler in routine care in our CHD unit of intensive care and anaesthesiology for cardiovascular surgery department.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Cerebral blood volume variation | at baseline
  Depending on stage of medico-surgical treatment
Cerebral blood volume variation | at baseline
  Depending on hemodynamic or ventilatory situation, and exposure to vasoactive or neuroactive drugs.

SECONDARY OUTCOMES:
Evolution of Arterial blood pressure | at baseline
Evolution of central venous blood pressure | at baseline
Evolution of left atrial pressure | at baseline
Evolution of SpO2 | at baseline
Evolution of SaO2 | at baseline
Evolution of SvO2 | at baseline
Evolution of PaCO2 | at baseline
Evolution of PaO2 | at baseline
Evolution of Hemoglobinemia | at baseline
Inotropic drugs dosages | at baseline
Vasopressive drugs dosages | at baseline
Sedation dosages | at baseline
Analgesia dosages | at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Haut Lévêque Cardiology Hospital, Pessac, France, France

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26472940/